CLINICAL TRIAL: NCT00690261
Title: The Impact of M1/M2 Tumor Associated Macrophage (TAM) Polarization on Cancer Progression and Prognosis Prediction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Chao-Chi Ho, National Taiwan University Hospital
Other Study IDs: 200709004R
Record Dates: First submitted 2008-06-01; First posted 2008-06-04 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-05

CONDITIONS: Tumor; Lung Cancer
Keywords: tumor associated macrophage; lung cancer; outcome
MeSH Terms: conditions — Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Pleural effusions and lung cancer tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- lung cancer: patients diagnosed of lung cancer with malignant pleural effusions

INTERVENTIONS:
Other:  — No intervention in this study
  Other Names: No intervention in this study

SUMMARY:
The purpose of this study is to evaluate the correlation between M1/M2 phenotype of tumor associated macrophage (TAM) in lung cancer patients and clinical outcome.

DETAILED DESCRIPTION:
Inflammatory response in the tumor micro-environment may facilitate the metastatic process (1). Macrophages are pivotal members of the inflammatory cells and the innate immune system within the tumor stroma. Tumor-associated macrophages can release growth factors, cytokines and inflammatory mediators that may facilitate cancer cell invasion, migration, angiogenesis, tumor progression or metastasis (1-5). A lot of studies showed TAM encounter factors that most frequently polarize them toward M2 type macrophage (1,4-5). It is interesting that in vitro studies macrophages have the potential to kill tumor by appropriate stimulation but these macrophage belonged to M1 and were not present in most tumor tissue (6). Some drugs target to suppress TAM have the promising results in animal models (7-9). Switching the TAM phenotype from M2 to M1 may promote anti-tumor activity (10). In this study we will correlate TAM M1/M2 ratio and patients' prognosis, the gene expression pattern of TAM.

References

1. Coussens LM, Werb Z. Inflammation and cancer. Nature 2002;420(6917):860-867.
2. Crowther M, Brown NJ, Bishop ET, Lewis CE. Microenvironmental influence on macrophage regulation of angiogenesis in wounds and malignant tumors. J Leukoc Biol 2001;70(4):478-490.
3. Lin EY, Nguyen AV, Russell RG, Pollard JW. Colony-stimulating Factor 1 Promotes Progression of Mammary Tumors to Malignancy. J. Exp. Med. 2001;193(6):727-740.
4. Mantovani A. Cancer Inflammation by remote control. Nature 2005;435(7043):752-753.
5. Pollard JW. Tumor-educated macrophages promote tumour progression and metastasis. Nature Reviews Cancer 2004;4(1):71-78.
6. Sica A, Schippa T, Mantovani A, Allavena P. Tumor-associated macrophage are distinct M2 polarized population promoting tumor progression: potential targets of anti-tumor therapy. Eur J of Cancer 2006;42:717-27
7. Sessa C, De Braud F, Perotti A, et al. Trabectedin for women with ovarian carcinoma after treatment with platinum and taxanes fails. J Clin Oncol 2005;23:1867-74.
8. Wahl L, Kleinman HK. Tumor-associated macrophages as targets for cancer therapy. J Natl Cancer Inst 1998;90:1583-4.
9. Giraudo E, Inoue M, Hanahan D. An amino-bisphosphonate targets MMP-9-expressing macrophages and angiogenesis to impair cervical carcinogenesis. J Clin Invest 2004;114:623-33.
10. Guiducci C, Vicari AP, Sangaletti S, Trinchieri G, Colombo MP. Redirecting in vivo elicited tumor infiltrating macrophages and dendritic cells towards tumor rejection. Cancer Res 2005;65:3437-46.

ELIGIBILITY:
Inclusion Criteria:

* lung cancer with malignant pleural effusions

Exclusion Criteria:

* None

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed of lung cancer with malignant pleural effusions
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-09; Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
outcome (treatment response and mortality) | 3 years

SECONDARY OUTCOMES:
clinical presentation | at enrollement

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Chi Ho, Principal Investigator — Department of Internal Medicine and Emergency Medicine, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan